CLINICAL TRIAL: NCT06102746
Title: A Single-center, Open Phase II Clinical Study of Surufatinib Plus Sintilimab Combined With Chemotherapy in the Treatment of Advanced Gastric Neuroendocrine Carcinoma
Brief Title: Clinical Study of Surufatinib Plus Sintilimab Combined With Chemotherapy in the Treatment of Advanced Gastric Neuroendocrine Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJMUCH-GI-GC03
Record Dates: First submitted 2023-10-18; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Gastric Neuroendocrine Carcinoma
Keywords: gastric neuroendocrine carcinoma; Sintilimab; Surufatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sintilimab + Surufatinib + EP: Sintilimab: 200mg intravenously administered on day 1; Surufatinib: 200mg/ day orally, taken continuously; Etoposide: 1, 2, 3 days of continuous administration, 100mg/m2, intravenous infusion; Cisplatin: 75mg/m2 on day 1, or 25mg/m2 on day 1, 2, and 3, intravenous infusion;
  Interventions: Drug: Sintilimab，Surufatinib

INTERVENTIONS:
Drug: Sintilimab，Surufatinib — Based on the standard EP regimen, the combination of surufatinib (anti-angiogenic therapy) and sintilimab (PD-1 inhibitor) were used among patients with advanced gastric neuroendocrine carcinoma.

SUMMARY:
This study aims to explore whether the combination of surufatinib (anti-angiogenic therapy) and sintilimab (PD-1 inhibitor) on the basis of EP regimen can further improve the effective rate and survival time of first-line treatment for patients with advanced gastric neuroendocrine carcinoma, and explore the safety and tolerability of this regimen.

DETAILED DESCRIPTION:
In this study, patients with advanced gastric neuroendocrine carcinoma were selected as the research object. Based on the standard EP regimen, the combination of surufatinib (anti-angiogenic therapy) and sintilimab (PD-1 inhibitor) could further improve the effective rate and survival time of patients, and explore the safety and tolerability of this treatment regimen.

Patients with advanced gastric neuroendocrine carcinoma who have not received systematic treatment will be treated with the following protocols:

Sintilimab: 200mg intravenously administered on day 1; Surufatinib: 200mg/ day orally, taken continuously; Etoposide: 1, 2, 3 days of continuous administration, 100mg/m2, intravenous infusion; Cisplatin: 75mg/m2 on day 1, or 25mg/m2 on day 1, 2, and 3, intravenous infusion; One treatment cycle every 21 days; Etoposide and cisplatin were used for a maximum of 4 cycles, after which maintenance therapy of solantinib and sindellizumab was administered, and the longest treatment cycle was 13 cycles (a total of 1 year). Patients received regular and periodic reviews, and imaging assessments were performed every 6 weeks after enrollment in the study. Safety will be evaluated by AE and laboratory tests. After disease progression, all patients were followed up with their secondary survival status every 3 months until death.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in this trial, patients must meet all of the following inclusion criteria:

1. Locally advanced or metastatic gastric neuroendocrine carcinoma (NEC), hyperproliferative neuroendocrine tumor (NET G3) or mixed neuroendocrino-non-neuroendocrine tumor (MiNEN), as demonstrated by pathology (WHO classification criteria 2019), may also be included;
2. Have not received systematic anti-tumor therapy before;
3. Have received radical treatment in the past and have no treatment interval from the end of chemotherapy, radiotherapy, or chemoradiotherapy to relapse for at least 6 months (the end time of the last chemotherapy cycle/the end time of the last radiotherapy);
4. There are measurable lesions defined by the RECIST 1.1 standard;
5. At least 18 years old;
6. ECOG physical condition: 0-1 score;
7. Expected survival of more than 3 months;
8. If the major organs function normally, the following criteria are met:

   1. Blood routine examination: hemoglobin (Hb) ≥90g/L; Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet (PLT) ≥100×10^9/L; White blood cell count (WBC) ≥3.0×10^9/L;
   2. Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (tumor liver metastasis, ≤5×ULN); Serum total bilirubin (TBIL) ≤1.5×ULN (Gilbert syndrome subjects, ≤3×ULN); Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥50ml/min;
   3. Coagulation function: activated partial thromboplastin time (APTT), International Standardized ratio (INR), prothrombin time (PT) ≤1.5×ULN;
9. The subjects voluntarily joined the study, signed the informed consent, and the compliance was good.

Exclusion Criteria:

Patients with any of the following conditions were excluded from the study:

1. The presence of a serious illness or medical condition, including but not limited to the following:

   1. Known recurrence in situ or metastasis at any other site;
   2. systemic active infection (i.e. infection resulting in body temperature ≥38 ° C);
   3. Clinically significant intestinal obstruction, pulmonary fibrosis, renal failure, liver failure, or symptomatic cerebrovascular disease;
   4. Severe/unstable angina, New York Heart Association (NYHA) Class III or IV symptomatic congestive heart failure;
   5. Clinically significant gastrointestinal bleeding;
   6. Known presence of human immunodeficiency virus (HIV) or acquired conventional immunodeficiency syndrome (AIDS) - associated disease, or active hepatitis B or C;
2. Pregnant or lactating women;
3. The researcher considers it inappropriate to enter this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First-line treatment for advanced gastric neuroendocrine carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  It refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including CR and PR cases. Solid tumor response assessment criteria (RECIST 1.1 criteria) were used to evaluate objective tumor response. Participants had to have a measurable tumor lesion at baseline, and response criteria were classified as complete response (CR), partial response (PR), stable disease (SD), and disease progression (PD) according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
PFS | 3 years
  From the date of enrollment to the date of the first onset of disease progression or death from any cause, whichever comes first. If the subject does not develop disease progression during the trial period, PFS is defined as the last date until the subject's last confirmed progression-free survival. Participants who discontinue the trial for reasons other than disease progression (no follow-up imaging) and those who receive post-trial treatment will be subject to data deletion based on the time of discontinuation or the time of initiation of post-trial treatment. When subjects do not use the time of discontinuation of the trial or the time of initiation of post-trial treatment as data deletion, pre-planned sensitivity statistical analyses will further confirm PFS based only on the time of the event at which image-confirmed progression occurs. New occurrence of other tumors is not considered a disease progression event and is not considered for data deletion. If the imaging examination

CONTACTS AND LOCATIONS:
Overall Officials: Ting Deng, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] 1.Dasari A, Shen C, Halperin D, Zhao B, Zhou S, Xu Y, et al. Trends in the Incidence, Prevalence,and Survival Outcomes in Patients With Neuroendocrine Tumors in the United States. JAMAOncol 2017;3:1335-1342 2.Leoncini E, Boffetta P, Shafir M, Aleksovska K, Boccia S, Rindi G. Increased incidence trendof low-grade and high-grade neuroendocrine neoplasms. Endocrine 2017;58:368-379 3.Nagtegaal ID, Odze RD, Klimstra D, Paradis V, Rugge M, Schirmacher P, et al. The 2019 WHOclassification of tumours of the digestive system. Histopathology 2020;76:182-188 4.Rindi G, Klimstra DS, Abedi-Ardekani B, Asa SL, Bosman FT, Brambilla E, et al. A commonclassification framework for neuroendocrine neoplasms: an International Agency for Research onCancer (IARC) and World Health Organization (WHO) expert consensus proposal. Mod Pathol2018;31:1770-1786 5.中国临床肿瘤学会神经内分泌肿瘤专家委员会. 中国胃肠胰神经内分泌肿瘤专家共识(2016年版). 临床肿瘤学杂志 2016;21:927-946 6.谭煌英, 娄彦妮, 罗杰, 刘继喜, 贾立群. 胃神经内分泌肿瘤的分型诊断和治疗. 中国医学前沿杂志：电子版 2014:5 7.Moertel CG, Kvols LK, O'Connell MJ, Rubin J. Treatment of neuroendocrine carcinomas withcombined etoposide and cisplatin. Evidence of major therapeutic activity in the anaplastic variantsof these neoplasms. Cancer 1991;68:227-232 8.Mitry E, Baudin E, Ducreux M, Sabourin JC, Rufié P, Aparicio T, et al. Treatment of poorlydifferentiated neuroendocrine tumours with etoposide and cisplatin. Br J Cancer 1999;81:1351-1355 9.Thomas KEH, Voros BA, Boudreaux JP, Thiagarajan R, Woltering EA, Ramirez RA. CurrentTreatment Options in Gastroenteropancreatic Neuroendocrine Carcinoma. Oncologist2019;24:1076-1088 10. Zhang P, Li J, Li J, Zhang X, Zhou J, Wang X, et al. Etoposide and cisplatin versusirinotecan and cisplatin as the first-line therapy for patients with advanced, poorly differentiatedgastroenteropancreatic neuroendocrine carcinoma: A randomized phase 2 study. Cancer 2020;126Suppl 9:2086-2092 11. Voron T, Colussi O, Marcheteau E, Pernot S, Nizard M, Pointet AL, et al. VEGF-A modulates expression of inhibitory checkpoints on CD8+ T cells in tumors. J Exp Med2015;212:139-148 12. Katoh M. FGFR inhibitors: Effects on cancer cells, tumor microenvironment and wholebody homeostasis (Review). Int J Mol Med2016;38:3-15 13. Xu J, Shen L, Bai C, Wang W, Li J, Yu X, et al. Surufatinib in advanced pancreaticneuroendocrine tumours (SANET-p): a randomised, double-blind, placebo-controlled, phase 3study. The Lancet Oncology 2020;21:1489-1499 14. Xu J, Shen L, Zhou Z, Li J, Bai C, Chi Y, et al. Surufatinib in advanced extrapancreaticneuroendocrine tumours (SANET-ep): a randomised, double-blind, placebo-controlled, phase 3study. The Lancet Oncology 2020;21:1500-1512